CLINICAL TRIAL: NCT02853045
Title: Comparison of Blood Pressure Control Achieved in Antihypertensive or Generic Drugs in Moderate to Severe Hypertensive Patients
Acronym: PRINGEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1408032; 2014-001404-22 (EudraCT Number)
Record Dates: First submitted 2016-07-06; First posted 2016-08-02 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Pharmaceutical Preparations; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- period with drug (trade name) then period with generic (Experimental): Period of 6 weeks.
  Interventions: Drug: period with drug (trade name) then period with generic
- period with generic then period with drug (trade name) (Experimental): Period of 6 weeks.
  Interventions: Drug: period with generic then period with drug (trade name)

INTERVENTIONS:
Drug: period with drug (trade name) then period with generic — The list of drugs is detailed in the "study description"
  Arms: period with drug (trade name) then period with generic
Drug: period with generic then period with drug (trade name) — The list of drugs is detailed in the "study description"
  Arms: period with generic then period with drug (trade name)

SUMMARY:
Despite a large diffusion for generic anti-hypertensive, they are not currently used.

Clinical validation studies could be better to convince users and prescribers than pharmacologic validation only.

A pragmatic study to evaluate generic anti-hypertensive efficacy is proposed. It takes place in real conditions of care for hypertensive patients, for a manometer control criteria.

The aim of the study is to test the hypothesis of non-inferiority for generic anti-hypertensive for blood pressure control.

DETAILED DESCRIPTION:
List of drugs : ALDACTONE, FLUMACH, SPIROCTAN, SPIRONONE, FLUDEX, INDATEN, LASILIX, TENSTATEN, ALDACTAZINE, PRINACTIZIDE, SPIROCTAZINE, MODURETIC, AVLOCARDYL, HEMIPRALON, STHASIN, BETATOP, TENORMINE, CELECTOL, DETENSIEL, FELSAN, KERLONE, RAGON, RONALOL, LOPRESSOR, SELOKEN, NEBILOX, TEMERIT, NEVEROL, SECTRAL, ACUITEL, KOREC, BRIEM, CIBACENE, COVERSYL, CAPTOLANE, LOPRIL, FOZITEC, ODRIK, GOPTEN, PRINIVIL, ZESTRIL, RENITEC, TEOULA, ZOFENIL, TRIATEC, KENOMON, ADALATE, CHRONOADALATE, AMLOR, BAYPRESS, DELTAZEN, DILRENE, DIACOR, MONO TILDIEM, FLODIL, IPERTEN, ISOPTINE, LERCAN, ZANIDIP, LEDELCARBERDIPE, LENIBERCARDIPE, DIBERLEPIDINE, XILERMIS, APROVEL, CRISARTERS, IFIRMASTA, FLUPPE, ZELMIRB, ATACAND, KENZEN, KARBIS, COZAAR, LOBERASNAT, LOTANBERSAR, MICARDIS, PRITOR, TOLURA, ZANACODAR, DINORTES, MIRPRESOC, NISIS, TAREG, CUENCA, TIFIVAL, VAGRECOR, VAMADRID, HYPERIUM, PHYSIOTENS, BIPRETERAX, PRETERAX, LODOZ, WYTENS, ACUILIX, KORETIC, BRIAZIDE, CIBADREX, CAPTEA, ECAZIDE, CORENITEC, ENALAVIS, ENALURETIC, COTRIATEC, RADOUCHE, FOZIRETIC, PRINZIDE, ZESTORETIC, COAPROVEL, IFIRMACOMBI, COCRISARTERS, COKENZEN, HYTACAND, COANHYVA, COHESAN , COTAREG, NISISCO, FORTZAAR, HYZAAR, MICARDISPLUS, PRITORPLUS, MARESSI, TOLUCOMBI, TENORDATE, BETA ADALATE

ELIGIBILITY:
Inclusion Criteria:

* hypertensive patient known and treated taking at least two antihypertensive
* Anti-hypertension treatment available in generic form
* Absence of changes in the anti-hypertension treatment during the previous 3 months

Exclusion Criteria:

* Patients on dialysis
* Patients with cardiac arrhythmia
* Patient refusing ambulatory blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Measure of systolic blood pressure | for 24 hours
  with holter (ambulatory)

SECONDARY OUTCOMES:
number of side effects | at 12 weeks
  number of side effects per patient with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MARIAT, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (8):
- France (8):
  - CH d'ANNONAY, Annonay
  - CH de FEURS, Feurs
  - CH de FIRMINY, Firminy
  - CH du PUY EN VELAY, Le Puy-en-Velay
  - CH de MONTBRISON, Montbrison
  - CH de ROANNE, Roanne
  - CH de SAINT-CHAMOND, Saint-Chamond
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No